CLINICAL TRIAL: NCT06951880
Title: A Phase I, Randomized, Single-blind, Placebo-controlled, 2-Part Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD4916 Following Single- and Multiple-ascending-dose Administration to Healthy Adult Volunteers (Including Japanese and Chinese Healthy Volunteers)
Brief Title: A Study to Investigate the Safety and Pharmacokinetics of Single- and Multiple-ascending Doses of AZD4916 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: D7340C00001
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: Single-ascending dose; Multiple-ascending dose; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD4916 (Experimental): Parts 1a and 2a participants will receive a single oral dose of AZD4916 on Day 1. Parts 1b and 2b participants will receive a single oral dose of AZD4916 on Day 1 and multiple doses of AZD4916 on Days 4 through 17.
  Interventions: Drug: AZD4916
- Placebo (Placebo Comparator): Parts 1a and 2a participants will receive a single oral dose of placebo on Day 1. Parts 1b and 2b participants will receive a single dose placebo on Day 1 and multiple doses of placebo on Days 4 through 17.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD4916 — AZD4916 will be administered as oral solution.
  Arms: AZD4916
Other: Placebo — Placebo will be administered as oral solution.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK) of AZD4916 in healthy adult participants.

DETAILED DESCRIPTION:
This is a single-blind, placebo-controlled study conducted at a single clinical unit.

The study will comprise of:

* Part 1: Single ascending dose (SAD) part (part 1a) and a Multiple ascending dose (MAD) part (part 1b), both in global participants.
* Part 2: SAD part (part 2a) and a MAD part (part 2b) specifically for Japanese and Chinese participants only.

ELIGIBILITY:
Main Inclusion Criteria:

* Healthy male and female participants with suitable veins for cannulation or repeated venipuncture.
* All females must have negative pregnancy test and females of childbearing potential must not be lactating and must agree to use an approved method of highly effective contraception.
* Have a Body Mass Index between 18 and 30 kg/m2 inclusive and weigh at least 45 kg at Screening.
* Part 2, Japanese participants only: Japanese participants must have been born in Japan, have 2 Japanese biological parents and 4 Japanese grandparents (as confirmed by the interview), and must not have lived outside of Japan for more than 10 years at the time of the Screening Visit.
* Part 2, Chinese participants only: Chinese participants must have been born in China (including Hong Kong, Macau, and Taiwan), have 2 Chinese biological parents and 4 Chinese grandparents (as confirmed by the interview), and must not have lived outside of China for more than 10 years at the time of the Screening Visit.

Main Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Principal Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of chest irradiation, fibrosis, malignancy, surgical procedure, trauma or liver disease.
* Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis results.
* Evidence of active tuberculosis or Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C virus (HCV) infection.
* Abnormal vital signs or clinically important abnormalities in rhythm.
* Current smokers, known or suspected history of alcohol, drug abuse or caffeine intake.
* History of severe allergy/hypersensitivity.
* Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* Participants who are vegans or have dietary restrictions.
* Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Estimated)
Dates: Start 2025-06-27 (Estimated); Primary Completion 2026-09-24 (Estimated); Study Completion 2026-09-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From Screening (Day -29 to Day -2) up to 44 days
  The safety and tolerability of AZD4916 following oral administration of single-ascending doses and multiple-ascending doses to healthy participants (including Japanese and Chinese) will be assessed.

SECONDARY OUTCOMES:
Area under concentration-time curve from time zero to infinity (AUCinf) | Part 1a and 2a: Up to Day 8, Part 1b and 2b: Up to Day 24
  The single-dose and steady-state PK of AZD4916 following oral administration of single-ascending doses and multiple-ascending doses of AZD4916 to healthy volunteers (including Japanese and Chinese healthy volunteers) will be characterised.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Part 1a and 2a: Up to Day 8, Part 1b and 2b: Up to Day 24
  The single-dose and steady-state PK of AZD4916 following oral administration of single-ascending doses and multiple-ascending doses of AZD4916 to healthy volunteers (including Japanese and Chinese healthy volunteers) will be characterised.
Area under concentration-time curve in the dosing interval (AUCtau) | Part 1a and 2a: Up to Day 8, Part 1b and 2b: Up to Day 24
  The single-dose and steady-state PK of AZD4916 following oral administration of single-ascending doses and multiple-ascending doses of AZD4916 to healthy volunteers (including Japanese and Chinese healthy volunteers) will be characterised.
Maximum observed drug concentration (Cmax) | Part 1a and 2a: Up to Day 8, Part 1b and 2b: Up to Day 24
  The single-dose and steady-state PK of AZD4916 following oral administration of single-ascending doses and multiple-ascending doses of AZD4916 to healthy volunteers (including Japanese and Chinese healthy volunteers) will be characterised.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/